CLINICAL TRIAL: NCT06955650
Title: First-in-man Imaging of a New PET Radiotracer for Oxytocin Receptors - Biodistribution and Radiation Dosimetry
Brief Title: First-in-man Imaging of a New PET Radiotracer for Oxytocin Receptors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Winterdahl, Associate professor in neuroimaging, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-004466-98
Record Dates: First submitted 2022-08-10; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pain, Face
Keywords: oxytocin; positron emission tomografi
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intranasal 13N-Oxytocin PET Imaging (Experimental): There is only one arm. All participants in the study will receive intranasal administration of a novel radiolabelled compound, 13N-Oxytocin, developed to selectively bind to oxytocin receptors. Following administration, participants will undergo positron emission tomography (PET) imaging to evaluate the in vivo distribution of the tracer, with a focus on uptake in the brain and trigeminal nerve regions.
  Interventions: Drug: Imaging procedure to measure the distribution of a newly developed radiolabeled ligand for the oxytocin receptor

INTERVENTIONS:
Drug: Imaging procedure to measure the distribution of a newly developed radiolabeled ligand for the oxytocin receptor — 13N-Oxytocin is a newly developed radiotracer designed to bind selectively to oxytocin receptors. It is labelled with nitrogen-13, a short-lived positron-emitting isotope, and is administered intranasally to facilitate direct access to the central nervous system via the nasal and trigeminal pathways. This radiotracer is investigational and is not intended to exert pharmacological effects. It is used solely for imaging purposes to assess the distribution and potential receptor binding sites of oxytocin in the human brain and the trigeminal nerve.
  Following administration, PET imaging is conducted using a hybrid PET/MRI scanner. The imaging procedure enables visualisation of the biodistribution of 13N-Oxytocin in vivo. The PET scan protocol includes dynamic image acquisition to track tracer uptake over time and is used in conjunction with MRI for precise anatomical localisation.

SUMMARY:
The investigators will test a new positron-emitting radiotracer to determine whether it is suitable for studying the oxytocin receptor by positron emission tomography (PET) in humans. If suitable, the radiotracer will be used to study the brain and trigeminal nerve in several disorders.

DETAILED DESCRIPTION:
The nine amino acid peptide oxytocin was first isolated in 1927 and is primarily recognised for its hormonal role in uterine contractions, lactation, and social bonding. It has been used to induce labour via infusion since the 1950s and was previously approved for nasal application to aid lactation, although its effectiveness for this purpose has since been questioned. Oxytocin is also involved in the modulation of pain within the body. It has been localised to the human dorsal root and trigeminal ganglia, and the terminals of hypothalamic neurons containing oxytocin-specific carrier proteins have been found in the dorsal horn of the spinal trigeminal nucleus. Oxytocin receptors have been identified in regions of the spinal cord associated with pain transmission in both non-human primates and rodents. Animal studies have provided evidence of oxytocin's analgesic effects, particularly following direct administration into the spinal canal or brain cavities.

Intrathecal administration of oxytocin, as opposed to intravenous delivery, has shown effectiveness in reducing chronic low back pain in humans, potentially involving the body's own opioid system. While direct access to the trigeminal system is challenging due to the skull's structure, a promising alternative is the nasocerebral pathway. This pathway enables certain substances administered nasally to reach central nervous system structures and has been explored as a method for delivering treatments to regions affected by neurodegenerative conditions.

Preliminary research suggests that intranasal delivery of oxytocin leads to pain relief restricted to areas supplied by the trigeminal nerve in both animals and humans. This effect appears to result from the nasal route enabling oxytocin to reach trigeminal receptors directly. In preclinical models, nasal but not systemic administration produced a significant analgesic effect in the face. Similar outcomes were observed in individuals with chronic migraine, where nasal oxytocin administration led to a strong reduction in facial pain. These findings suggest that intranasal oxytocin may work by concentrating in the trigeminal nerve via the nasocerebral route.

The current study aims to evaluate how oxytocin distributed via nasal administration spreads in the body, using positron emission tomography (PET). This imaging technique will allow visualisation of how the compound moves through the body and whether it reaches relevant structures such as the trigeminal nerve. The goal is to better understand how intranasal oxytocin might enable targeted pain relief and potentially support its use in treating conditions related to the trigeminal system.

ELIGIBILITY:
Inclusion Criteria:

* Female or male age 35-50 (Women of childbearing potential must use birth control and test negative for pregnancy prior to enrollment in this study).
* Normal anatomy in nasal region evaluated with MRI
* Normal sensory function evaluated with "The Sniffin' Sticks Olfactory Test-Kits

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Metal implanted in the body.
* Diseases of the nose and airways.
* Former or current cancer in the head/neck area where radiation therapy was applied.
* Former or current brain disease.
* Psychiatric diseases.
* Heart disease.
* Other serious chronic or acute disease.
* Substance abuse disorders.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Radiation dosimetry of 13N-Oxytocin calculated using MIRDcalc | Up to 14 days post-administration
  Description: Radiation dosimetry will be calculated based on dynamic PET scan data using MIRDcalc software. Organ-specific absorbed radiation doses and effective dose will be reported based on ICRP Publication 103 guidelines.
  Units of Measure: Millisievert (mSv), milligray (mGy)

SECONDARY OUTCOMES:
Biodistribution of 13N-Oxytocin assessed by PET imaging | Up to 14 days post-administration
  Description: The biodistribution of 13N-Oxytocin will be assessed using PET imaging in combination with MRI for anatomical localisation. Standardised Uptake Values (SUVs) will be calculated using PMOD software to quantify tracer uptake in predefined brain regions and the trigeminal nerve.
  Units of Measure: Standardised Uptake Value (SUV)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Winterdahl M, Nielsen EN, Hansen SB, Dias AH, Vendelbo MH, Jakobsen S, Yeomans D. First-in-human intranasal [13N]oxytocin PET: evaluation of feasibility, biodistribution, and radiation dosimetry. EJNMMI Res. 2025 Nov 18;15(1):137. doi: 10.1186/s13550-025-01329-0. PMID 41251983